CLINICAL TRIAL: NCT01886066
Title: Accuracy of Sentinel Lymph Node Biopsy in Nodal Staging of High Risk Endometrial Cancer: A Prospective Trial
Brief Title: Accuracy of Sentinel Lymph Node Biopsy in Nodal Staging of High Risk Endometrial Cancer
Acronym: EndoSLN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0257-C
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node; Indocyanine Green
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This is an Investigator-Initiated Prospective Trial (not a clinical trial, as ICG not a novel drug that is being used as intervention).

ARMS (1):
- Indocyanine Green (Experimental): All patients on study will have ICG injection for SLN mapping
  Interventions: Biological: Indocyanine Green (ICG)

INTERVENTIONS:
Biological: Indocyanine Green (ICG) — ICG (Indocyanine Green) will be used as a fluorescent agent to identify sentinel lymph nodes intraoperatively. One 25 mg vial of ICG will be reconstituted in 10 mL of aqueous solvent (2.5 mg/mL). The solution will be injected at the 3 and 9 o'clock positions of the cervical stroma. 0.5 mL is injected superficially (submucosa) and 0.5 mL is injected deep (~8mm) in the cervical stroma for a total injection volume of 2 mL.

SUMMARY:
The standard of care for women with high risk endometrial cancer is the removal of all visible lymph nodes in the pelvis and lower abdomen to identify if disease has spread to these areas. It is estimated that no more than 25% of all women with presumed early stage high risk endometrial cancer will have positive lymph nodes however currently the majority of women are subjected to extensive resection of all pelvic lymph and or para-aortic lymph nodes and its associated morbidities. The objective of this study is to determine if intraoperative sentinel lymph node (SLN) mapping will improve the assessment of regional lymph nodes and enhance the detection of lymph nodes with metastatic disease in endometrial cancer. This would benefit the majority of women with early stage high risk endometrial cancer and would prevent the associated complications of pelvic lymph node dissection.

DETAILED DESCRIPTION:
If the SLN can be accurately identified and the detection of metastatic lymph nodes in women with early stage high risk endometrial cancer can be improved then the majority of women could avoid a complete systematic pelvic lymphadenectomy. Pelvic lymphadenectomy is associated with many intraoperative and postoperative complications such as hemorrhage, lymphocyst formation, nerve injury and chronic lower extremity lymphedema. If less invasive techniques to assess regional lymph node involvement, such as SLN mapping, replaced routine pelvic lymphadenectomy the complications associated with more extensive pelvic surgery could be avoided.

This will be a prospective cohort study. The population to be studied will be patients with newly diagnosed early stage high risk endometrial cancer who will undergo primary surgical intervention that includes hysterectomy and bilateral pelvic and inframesenteric para-aortic lymphadenectomy via laparotomy, laparoscopy or robotic-assisted. Patients will be taken to the operating room for their planned procedure. After initiation of general anesthesia, fluorescent dye (indocyanine green, ICG) will be injected into the patient's cervix. The dye will be visualized by excitation with an infrared light (an attachment on the Novadaq Pinpoint system for laparoscopy). The surgery will proceed and all lymph nodes that are "green" will be removed surgically and their anatomic location and laterality documented. These "green" sentinel nodes will be assessed by a study pathologist by frozen section and the result read out intraoperatively. The hysterectomy and complete lymphadenectomy will then be performed. The SLN status will be compared to the status of the other nodes removed at complete lymphadenectomy. All data on these patients will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrial cancer with high risk histologic subtypes including grade 3 endometrioid, carcinosarcoma, serous, clear cell, undifferentiated adenocarcinoma, and and any mixed high risk histology.
* Clinical stage 1 disease- no evidence of metastatic disease beyond the uterus by physical exam or preoperative imaging if performed.
* Patients who have signed an approved informed consent.
* Patients who will undergo surgery that includes a hysterectomy and bilateral pelvic and inframesenteric para-aortic lymphadenectomy via laparoscopy or robotic-assisted.

Exclusion Criteria:

* Women with grade 1 or 2 endometrioid adenocarcinoma
* Patients with evidence of metastatic disease on preoperative imaging.
* Patients with evidence of intraperitoneal metastatic disease intraoperatively (patients with suspicious retroperitoneal lymph nodes intraoperatively will still be included).
* Patients with known allergy to iodine compounds
* Pregnant patient.
* Patients with previous retroperitoneal surgery.
* Patients with previous history of pelvic/abdominal radiation.
* Patients with recurrent endometrial cancer.
* Any patient treated with neoadjuvant chemotherapy and/or radiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-03; Primary Completion 2019-06-21 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Performance Analysis | Year 3
  Performance analyses of SLN mapping will be performed. In particular, sensitivity, specificity, and predictive accuracy of mapping and detection of sentinel lymph nodes with metastatic disease will be calculated using the pathology results of the surgical intervention as the Standard of Reference. Performance analyses will be evaluated at both the lesion and patient level. Generalized estimating equations will be used to adjust for correlations of repeated measures within patients. Raw performance estimates will be reported with adjusted 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ferguson, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Marchocki Z, Cusimano MC, Vicus D, Pulman K, Rouzbahman M, Mirkovic J, Cesari M, Maganti M, Zia A, Ene G, Ferguson SE. Diagnostic accuracy of frozen section and patterns of nodal spread in high grade endometrial cancer: A secondary outcome of the SENTOR prospective cohort study. Gynecol Oncol. 2023 Jun;173:41-48. doi: 10.1016/j.ygyno.2023.04.004. Epub 2023 Apr 18. PMID 37075495